CLINICAL TRIAL: NCT05480098
Title: Efficacy of Intraoperative Brimonidine for Hemostasis During Eyelid Surgery
Brief Title: Brimonidine for Intraoperative Hemostasis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Fellow graduated prior to enrollment
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Christopher James Compton, Associate Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21.0989
Record Dates: First submitted 2022-06-06; First posted 2022-07-29 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Dermatochalasis of Eyelid; Ptosis, Eyelid; Ectropion; Entropion
MeSH Terms: conditions — Blepharoptosis; Ectropion; Entropion | interventions — Brimonidine Tartrate

STUDY DESIGN:
Intervention Model Description: A randomized, prospective clinical trial will be performed with IRB approval to compare intraoperative application of ophthalmic brimonidine solution to standard methods of hemostasis control. This study will be blinded to the surgeon grading the severity of bleeding and the patient unaware which side would receive the intervention. Topical brimonidine ophthalmic solution will be placed intraoperatively to the open surgical wound of one eyelid and we will assess the severity of bleeding via a surgeon's grading scale. The fellow eye's surgical wound will be used as the control. The laterality of intervention is randomized. Reduction of bleeding severity is the primary outcome as graded by a subjective surgeon's grading scale. A secondary outcome may be severity of postoperative bruising in the study eye versus the fellow control eye, as graded by post-operative bruising severity.
Who Masked: Participant, Care Provider
Masking Description: This study will be blinded to the surgeon grading the severity of bleeding and the patient will be unaware which side would receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brimonidine intervention (Experimental): We will compare hemostasis between 2 surgical sides of the same patient. One side will be randomized to receive Brimonidine (0.15% or 0.2%) in addition to standard hemostasis measures, while the other side will receive only standard hemostasis measures (preoperative discontinuation of blood thinners, preoperative injection of lidocaine with epinephrine).
  Interventions: Drug: Brimonidine Topical
- Control Arm (No Intervention): We will compare hemostasis between 2 surgical sides of the same patient. One side will be randomized to receive Brimonidine (0.15% or 0.2%) in addition to standard hemostasis measures, while the other side will receive only standard hemostasis measures (preoperative discontinuation of blood thinners, preoperative injection of lidocaine with epinephrine).

INTERVENTIONS:
Drug: Brimonidine Topical — Topical brimonidine intraoperatively for hemostasis
  Other Names: Alphagan
  Arms: Brimonidine intervention

SUMMARY:
The purpose of this study is to observe and report the effects of topical ophthalmic brimonidine in oculofacial plastic surgery.

DETAILED DESCRIPTION:
Brimonidine ophthalmic solution (Alphagan) is mainstay in glaucoma therapy to reduce intraocular pressure. The medication is an alpha2 adrenergic agonist, which increases uveoscleral outflow of aqueous humor. Alpha2 agonists also have vasoconstrictive properties, which has been utilized in over-the-counter medications like Lumify for redness relief. An unexploited utility of its vasoconstrictive property is reduction in intraoperative bleeding during ophthalmic surgery. The purpose of this study is to observe and report the effects of brimonidine in oculofacial plastic surgery.

There are reports in ophthalmic literature that observe the hemostatic effect of topical brimonidine across different subspecialties. It has been shown to reduce intraoperative bleeding and post-operative subconjunctival hemorrhages in pterygium removal, strabismus surgery, LASIK, and cataract surgery. One study claimed that it had a comparable hemostatic effect to phenylephrine.

Many of the procedures in oculoplastic surgery involve manipulation and incision of eyelid skin and conjunctival tissue. Some examples include blepharoplasty, ptosis repair, medial spindles, lateral tarsal strips, canthotomy and cantholysis with subsequent repair, retraction repair, and orbital fracture repair. Rapid and adequate control of intraoperative bleeding is crucial to the success of oculoplastic surgery. Although surgeons take proper precautions to prevent inadequate hemostasis (discontinuing blood thinners, use of electrocautery, and administration of intradermal epinephrine), excessive bleeding can still occur. This can impair surgeon performance by obscuring visualization, and negatively affect the patient due to prolonged operative times, and delayed healing due to hematoma formation. The most feared complication of oculoplastic surgery is intraorbital hemorrhage, which can cause orbital compartment syndrome causing vision loss.

Therefore, any intervention to minimize bleeding is very advantageous to the patient. Use of Brimonidine drops intraoperatively will improve hemostasis, resulting in improved visualization, reduced operative time under anesthesia, and reduced risk of significant intraorbital hemorrhage. Due to both brimonidine's vasoconstrictive properties and relatively favorable safety profile, it raises the question: can brimonidine be used to achieve better hemostasis in oculoplastic procedures?

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 18
* Ophthalmic conditions requiring oculoplastic surgery

Exclusion Criteria:

* Known allergy or adverse effects to brimonidine
* Hypotony
* Acute ophthalmic infection
* History of hypotension
* Orthostatic hypotension
* Pregnancy
* History of Central Nervous System (CNS) depression from medication use
* Thrombotic disorders
* Asymmetrical oculoplastic conditions that may interfere with tear drainage (e.g. unilateral NLDO)
* Current use of brimonidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Hemostasis | At the time of surgery.
  Change in Hemostasis Score

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Compton, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hong S, Kim CY, Seong GJ, Han SH. Effect of prophylactic brimonidine instillation on bleeding during strabismus surgery in adults. Am J Ophthalmol. 2007 Sep;144(3):469-70. doi: 10.1016/j.ajo.2007.04.038. PMID 17765438
- [Background] Ucar F, Cetinkaya S. The Results of Preoperative Topical Brimonidine Usage in Pterygium Surgery. J Ocul Pharmacol Ther. 2020 May;36(4):234-237. doi: 10.1089/jop.2019.0085. Epub 2020 Feb 27. PMID 32105500
- [Background] Kim DH, Yang HK, Han SB, Hwang JM. Effect of Topical Brimonidine 0.15% on Conjunctival Injection after Strabismus Surgery in Children. J Ophthalmol. 2021 May 4;2021:5574194. doi: 10.1155/2021/5574194. eCollection 2021. PMID 34055396
- [Background] Kim CS, Nam KY, Kim JY. Effect of prophylactic topical brimonidine (0.15%) administration on the development of subconjunctival hemorrhage after intravitreal injection. Retina. 2011 Feb;31(2):389-92. doi: 10.1097/IAE.0b013e3181eef28e. PMID 20890238
- [Background] Ucar F, Cetinkaya S. The Results of Preoperative Use of Topical Brimonidine in Strabismus Surgery. J Ocul Pharmacol Ther. 2021 May;37(4):230-235. doi: 10.1089/jop.2020.0144. Epub 2021 Mar 8. PMID 33684337